CLINICAL TRIAL: NCT06972680
Title: Determination of the Optimal Volume of 0.5% Bupivacaine Liposome in Single-Injection Interscalene Brachial Plexus Block: A Bayesian Phase I/II Trial
Status: Enrolling by invitation | Type: Observational
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Affiliated Hospital of Jiaxing University, Affiliated Hospital of Jiaxing University
Other Study IDs: 2025-LP-076
Record Dates: First submitted 2025-04-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Arthroscopy
Keywords: Interscalene brachial plexus block; Phrenic nerve block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Interscalene brachial plexus block
  Interventions: Drug: Bupivacaine Liposomes(BL)

INTERVENTIONS:
Drug: Bupivacaine Liposomes(BL) — Prior to surgery, an interscalene brachial plexus block was performed, injecting the preset volume of 0.5% bupivacaine liposomes according to the Bayesian optimal interval method.

SUMMARY:
This single-center, prospective, single-arm, Bayesian phase I/II clinical trial evaluates the incidence of HDP following ISB in shoulder arthroscopy and determines the optimal volume of a single injection of liposomal bupivacaine.

DETAILED DESCRIPTION:
Based on the ISB being the optimal nerve block for post-arthroscopic shoulder surgery analgesia and the potent analgesic effect of bupivacaine liposomes, this study aims to explore the optimal volume of a single ISB injection of bupivacaine liposomes in shoulder arthroscopy using the Bayesian Optimal Interval Design, with the goal of achieving the same analgesic effect while minimizing the incidence and duration of HDP to the greatest extent.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above;
* ASA classification I-III;
* Undergoing arthroscopic rotator cuff repair, capsular tightening, acromioplasty, synovectomy,.

Exclusion Criteria:

* History of pulmonary disease;
* Abnormal coagulation function or coagulation disorders;
* History of local anesthetic allergy;
* Infection, lesion, or history of cervical disease at the block site;
* Pregnancy;
* Refusal to participate in the study or inability to communicate;
* Long-term use of opioids;
* Body mass index >35 kg/m2;
* History of nerve injury, paralysis, or paresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective arthroscopic shoulder surgery at Jiaxing University Affiliated Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Hemidiaphragmatic paresis incidence rate(Phase Ⅰ) | Perioperative
  The diaphragmatic excursion was measured using ultrasound 0.5 hours after the completion of the nerve block, and partial or complete unilateral Hemidiaphragmatic paresis(HDP) was assessed based on the diaphragmatic excursion. No excursion was defined as ≤25%, partial excursion as >25% and ≤75%, and complete excursion as >75%. A diaphragmatic excursion greater than or equal to 25% measured by ultrasound can be defined as HDP.
Success rate of interscalene brachial plexus block (Phase II) | Perioperative
  Before the surgery, an ultrasound-guided interscalene brachial plexus block is performed. After the surgery, when the patient is fully awake, a simplified sensory-motor assessment scale is used for evaluation. A comprehensive score of ≥12 is defined as a successful nerve block.

SECONDARY OUTCOMES:
Hemidiaphragmatic paresis incidence rate | Perioperative
  The diaphragmatic excursion was measured using ultrasound 6 hours and 24 hours after the completion of the nerve block, and partial or complete unilateral Hemidiaphragmatic paresis(HDP) was assessed based on the diaphragmatic excursion. No excursion was defined as ≤25%, partial excursion as >25% and ≤75%, and complete excursion as >75%. A diaphragmatic excursion greater than or equal to 25% measured by ultrasound can be defined as HDP.
Lung function | Perioperative
  Lung function parameters, including tidal volume, vital capacity, and forced vital capacity, were measured bedside using a portable respiratory function monitor at 0.5 hours, 6 hours, and 24 hours after nerve block.

CONTACTS AND LOCATIONS:
Overall Officials: Mingzi An, MD, Principal Investigator — Jiaxing University Affiliated Hospital
Locations (1):
- Jiaxing University Affiliated Hospital, Jiaxing, Zhejiang, China